CLINICAL TRIAL: NCT01627132
Title: Discontinuation of Dasatinib in Patients With Chronic Myeloid Leukemia in Chronic Phase Who Have Maintained Complete Molecular Remission for Two Years; Dasatinib Stop Trial
Brief Title: Discontinuation of Dasatinib in Patients With Chronic Myeloid Leukemia-CP Who Have Maintained Complete Molecular Remission for Two Years; Dasatinib Stop Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shimousa Hematology Study Group (Other)
Collaborators: Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Principal Investigator, Koiti Inokuchi,MD,PhD., Nippon Medical School, Shimousa Hematology Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSG-01
Record Dates: First submitted 2012-02-14; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dasatinib (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 100mg QD
  Other Names: BMS-354825

SUMMARY:
The purpose of this study is to assess whether dasatinib can be discontinued without occurrence of molecular relapse in patients with chronic myeloid leukemia in chronic phase in complete molecular remission (CMR) while on dasatinib.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Myeloid Leukemia in the Chronic Phase.
* Patients with BCR-ABL-negative checks.
* 15 years old over.
* ECOG performance status (PS) score 0-2.
* Adequate organ function (hepatic, renal and lung).
* Signed written informed consent.

Exclusion Criteria:

* A case with the double cancer of the activity.
* Women who are pregnant or breastfeeding.
* Patients with complications or a history of severe.
* Patients with mutation of T315I、F317L、V299L.
* Patients with additional chromosome abnormalities.
* The case of Pleural effusion with poor control.
* Patients with a history of hematopoietic stem cell transplantation.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-02 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The overall probability of maintenance of complete molecular remission at 12 months after stopping dasatinib. | at 12 months

SECONDARY OUTCOMES:
Rate of complete molecular remission that will be sustained after dasatinib rechallenge. | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Koiti Inokuchi, Principal Investigator — Nippon Medical School
Locations (1):
- Nippon Medical School, Sendagi 1-1-5, Bunkyo-ku,Tokyo, Japan

REFERENCES:
- [Derived] Kumagai T, Nakaseko C, Nishiwaki K, Yoshida C, Ohashi K, Takezako N, Takano H, Kouzai Y, Murase T, Matsue K, Morita S, Sakamoto J, Wakita H, Sakamaki H, Inokuchi K; Kanto CML, Shimousa Hematology Study Groups. Silent NK/T cell reactions to dasatinib during sustained deep molecular response before cessation are associated with longer treatment-free remission. Cancer Sci. 2020 Aug;111(8):2923-2934. doi: 10.1111/cas.14518. Epub 2020 Jun 26. PMID 32614159